CLINICAL TRIAL: NCT04136041
Title: Study Protocol for a Pilot Randomized Controlled Trial on a Smartphone Application-based Intervention for Subthreshold Depression
Brief Title: Study Protocol for a Smartphone Application-based Intervention for Subthreshold Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kibi International University (Other)
Responsible Party: Principal Investigator, Kazuki Hirao, PhD, OT, Assistant Professor, Kibi International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-33
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Subthreshold Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone Application (Experimental): Participants watch a video using the Smartphone Application displaying positive word stimuli.
  Interventions: Device: Smartphone Application
- No Intervention (No Intervention): No Intervention.

INTERVENTIONS:
Device: Smartphone Application — The experimental group will watch movies using the Smartphone application for at least 10 min a day for 5 weeks.
  Arms: Smartphone Application

SUMMARY:
The investigators plan to conduct a randomized controlled trial to examine whether a Smartphone-based Intervention improves subthreshold depression symptoms compared to no intervention.

The purpose of this pilot randomized controlled trial is to investigate the feasibility of the final randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* Males and females
* Center for Epidemiologic Studies Depression Scale score ≥16
* Written informed consent prior to participation
* Owns a smartphone with the iOS® operating system

Exclusion Criteria:

* Lifetime history of psychiatric disorders
* Currently receiving treatment for a mental health problem from a mental health professional
* Experience of a major depressive episode in the 2 weeks prior to the study, as ascertained using the Mini-International Neuropsychiatric Interview
* Vision or hearing deficits that negatively impact everyday life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Depression severity as measured by the Center for Epidemiologic Studies Depression Scale (CES-D) score. | Change from Baseline CES-D at 5 weeks
  The CES-D is a 20-item self-report questionnaire used to measure depressive symptoms. The CES-D is a four-point Likert scale, with each item scored from 0 to 3. The total score ranges from 0 to 60 points. The higher the score, the stronger the depressive symptoms.

SECONDARY OUTCOMES:
Psychological distress as measured by the Kessler Screening Scale for Psychological Distress (K6) score. | Change from Baseline K6 at 5 weeks
  The K6 is a 6-item self-report questionnaire used to measure psychological distress. The K6 is a five-point Likert scale, with each item scored from 0 to 4. The total score ranges from 0 to 24 points. The higher the score, the stronger the psychological distress.
Anxiety as measured by the 7-item Generalized Anxiety Disorder Scale (GAD-7). | Change from Baseline GAD-7 at 5 weeks
  The GAD-7 is a 7-item self-report questionnaire used to measure anxiety. The GAD-7 is a four-point Likert scale, with each item scored from 0 to 3. The total score ranges from 0 to 21 points. The higher the score, the stronger the anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Kibi International University, Takahashi, Okayama-ken, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kato Y, Kageyama K, Mesaki T, Uchida H, Sejima Y, Marume R, Takahashi K, Hirao K. Study protocol for a pilot randomized controlled trial on a smartphone application-based intervention for subthreshold depression: Study protocol clinical trial (SPIRIT Compliant). Medicine (Baltimore). 2020 Jan;99(4):e18934. doi: 10.1097/MD.0000000000018934. PMID 31977910